CLINICAL TRIAL: NCT04248465
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multicenter Study With an Open-Label Extension to Evaluate the Efficacy and Safety of Ravulizumab in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: An Efficacy and Safety Study of Ravulizumab in ALS Participants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The IDMC recommended the study be discontinued due to lack of efficacy with ravulizumab.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN1210-ALS-308; 2019-004619-30 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: Ravulizumab; ALXN1210; Ultomiris; Motor Neuron Disease; Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental): Participants will receive ravulizumab for the duration of the study.
  Interventions: Biological: Ravulizumab
- Placebo (Placebo Comparator): Participants will receive placebo during the 50-week Randomized Controlled Period of the study, after which they will enter the Open-label Extension Period of the study and switch to receive ravulizumab.
  Interventions: Drug: Placebo; Biological: Ravulizumab

INTERVENTIONS:
Drug: Placebo — Single loading dose via intravenous infusion, followed by regular maintenance dosing, based on weight.
  Arms: Placebo
Biological: Ravulizumab — Single loading dose via intravenous infusion, followed by regular maintenance dosing, based on weight.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The purpose of the study is to assess the efficacy and safety of ravulizumab for the treatment of adult participants with ALS.

ELIGIBILITY:
Key Inclusion Criteria:

1. A diagnosis of sporadic or familial ALS, defined by the El Escorial criteria (possible, laboratory-supported probable, probable, or definite ALS).
2. ALS onset ≤ 36 months from Screening.
3. Documented meningococcal vaccination not more than 3 years prior to, or at the time of, initiating study treatment.
4. Upright slow vital capacity ≥ 65% predicted at Screening.
5. If on riluzole, participant must be on a stable dose for 30 days; if on edaravone, participant must be on a stable dose for 60 days (2 cycles).
6. Body weight ≥ 40 kilograms at Screening.
7. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Key Exclusion Criteria:

1. History of Neisseria meningitidis infection.
2. Human immunodeficiency virus (HIV) infection (evidenced by HIV 1 or HIV 2 antibody titer).
3. Dependence on invasive or non-invasive mechanical ventilation.
4. Previously or currently treated with a complement inhibitor.
5. Exposure to an investigational drug or device within 30 days of Screening or 5 half lives of the study drug, whichever is greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (34):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Neuromuscular Research Center and Clinic, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - University of California-Irvine, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - University of California San Diego Medical Center, San Diego, California
  - Norris MDA/ALS Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus School of Medicine, Aurora, Colorado
  - University of Florida at Shands Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Las Vegas Clinic, Las Vegas, Nevada
  - Beth Israel Medical Center - PRIME, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Atrium Health Neuroscience Institute, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - Houston Methodist Neurological Institute-Movement Disorders Clinic, Houston, Texas
  - Nerve & Muscle Center of Texas, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Neurology Clinical and Translational Research Office, Richmond, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
- Australia (4):
  - Brain and Mind Centre, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- UZ Leuven, Leuven, Belgium
- Canada (7):
  - Heritage Medical Research Centre (HMRC), Edmonton, Alberta
  - Stan Cassidy Center for Rehabilitation, Fredericton, New Brunswick
  - LHSC - University Hospital, London, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - University Hospital of Quebec-Universite Laval, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Denmark (3):
  - Ålborg Universitets Hospital, Aalborg
  - Aarhus University Hospital Department of Neurology, Aarhus
  - Bispebjerg Hospital, Copenhagen
- France (8):
  - CHU de Nice Hôpital Pasteur 2, Nice, Alpes Maritimes
  - CHU de Limoges - Hôpital Dupuytren, Limoges, Haute Vienne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Tours - Hôpital Bretonneau, Tours, Indre Et Loire
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - Hopital Roger Salengro - CHU Lille, Lille
  - Hôpital de la Timone, Marseille
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (5):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Universitaetsmedizin Goettingen, Goettigen, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Jena, Jena, Thuringia
- Beaumont Hospital, Dublin, Ireland
- Israel (3):
  - Rambam Health Care Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Ospedale San Raffaele, Milan
  - ICS Maugeri IRCCS, Milan
  - Istituto Auxologico Italiano, Milan
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale Civile di Baggiovara, Modena
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - University of Turin, Torino
- Japan (10):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - Yoshino Neurology Clinic, Ichikawa-shi, Chiba
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokushima University Hospital, Tokushima, Tokushima
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City, Tokyo-To
  - Toho University Omori Medical Center, Ōta-ku, Tokyo-To
  - Keio University Hospital, Shinjuku-Ku, Tokyo-To
- University Medical Centre Utrecht, Utrecht, Netherlands
- CityClinic, Warsaw, Poland
- Spain (5):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Rafael, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Karolinska Trial Alliance (KTA), Huddinge
  - Norrlands universitetssjukhus, Umeå
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- United Kingdom (2):
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Royal Hallamshire Hospital, Sheffield, West Midlands

REFERENCES:
- [Derived] Genge A, van den Berg LH, Frick G, Han S, Abikoff C, Simmons A, Lin Q, Patra K, Kupperman E, Berry JD. Efficacy and Safety of Ravulizumab, a Complement C5 Inhibitor, in Adults With Amyotrophic Lateral Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2023 Oct 1;80(10):1089-1097. doi: 10.1001/jamaneurol.2023.2851. PMID 37695623

RESULTS

PARTICIPANT FLOW:
Groups:
- Ravulizumab/Ravulizumab: Participants received a weight-based loading dose of ravulizumab on Day 1, followed by a weight-based maintenance dose on Day 15, then once every 8 weeks (q8w) up to Week 42 (inclusive) during the Randomized Controlled Period. Then during the Open Label Extension Period, participants received ravulizumab, with a blinded 900 milligrams (mg) dose at Week 50, followed by an open-label ravulizumab maintenance dose at Week 52, then q8w for up to 106 weeks of treatment.
- Placebo/Ravulizumab: Participants received a weight-based loading dose of placebo matched to ravulizumab on Day 1, followed by a weight-based maintenance dose on Day 15, then q8w up to Week 42 (inclusive) during the Randomized Controlled Period. Then during the Open Label Extension Period, participants received ravulizumab, with a blinded loading dose at Week 50, followed by an open-label ravulizumab maintenance dose at Week 52, then q8w for up to 106 weeks of treatment.
Period: Randomized-Controlled Period
Arm/Group | Ravulizumab/Ravulizumab | Placebo/Ravulizumab
Started | 255 | 127
Received at Least 1 Dose of Study Drug | 255 | 127
Completed | 15 | 5
Not Completed | 240 | 122
Not completed — Death | 12 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Study Terminated by Sponsor | 194 | 99
Not completed — Withdrawal by Subject | 30 | 17
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Open-label Extension Period
Arm/Group | Ravulizumab/Ravulizumab | Placebo/Ravulizumab
Started | 14 | 5
Received at Least 1 Dose of Study Drug | 14 | 5
Completed | 0 | 0
Not Completed | 14 | 5
Not completed — Study Terminated by Sponsor | 14 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug grouped by randomized treatment group.
Groups:
- Ravulizumab: Participants received a weight-based loading dose of ravulizumab on Day 1, followed by a weight-based maintenance dose on Day 15, then q8w up to Week 42 (inclusive) during the Randomized Controlled Period. Then, during the Open Label Extension Period, participants received ravulizumab, with a blinded 900 mg dose at Week 50, followed by an open-label ravulizumab maintenance dose at Week 52, then q8w for up to 106 weeks of treatment.
- Placebo: Participants received a weight-based loading dose of placebo matched to ravulizumab on Day 1, followed by a weight-based maintenance dose on Day 15, then q8w up to Week 42 (inclusive) during the Randomized Controlled Period. Then during the Open Label Extension Period, participants received ravulizumab, with a blinded loading dose at Week 50, followed by an open-label ravulizumab maintenance dose at Week 52, then q8w for up to 106 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | Ravulizumab | Placebo | Total
Number analyzed (Participants) | 255 | 127 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.57) | 58.0 (11.03) | 58.4 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 58 | 152
  Male | 161 | 69 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 12 | 34
  Not Hispanic or Latino | 205 | 105 | 310
  Unknown or Not Reported | 28 | 10 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 22 | 12 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 202 | 103 | 305
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 26 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Total Score
Description: The ALSFRS-Revised is a validated instrument for evaluating the levels of the functional status of participants with amyotrophic lateral sclerosis (ALS) in 4 areas, including bulbar, gross motor activity, fine motor activity, and respiratory functions. The scale included 12 functional items and each item is rated on a 0 to 4 scale, with a maximum total score of 48. A higher score indicated greater retention of function. Baseline was defined as last non-missing value on or before first study drug administration.
Time Frame: Baseline, Week 50
Population: FAS included all randomized participants who received at least 1 dose of study drug grouped by randomized treatment group. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 32 | 14
units on a scale | -11.9 (7.30) | -10.6 (6.05)

2. Secondary Outcome: Time To Ventilator Assistance-free Survival
Description: Ventilation Assistance-Free Survival (VAFS) is a composite endpoint of survival and severe and irreversible respiratory decline. The use of VAFS allowed for the collection of survival data that was not impacted by survival prolongation from noninvasive or permanent ventilatory interventions which could prolong life without impacting underlying disease progression.
Time Frame: Up to Week 50
Population: FAS included all randomized participants who received at least 1 dose of study drug grouped by randomized treatment group.
Measure: Median (Full Range); unit: months
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 255 | 127
months | 6.05 [0.79 to 11.10] | 7.69 [4.83 to 9.53]

3. Secondary Outcome: Change From Baseline In Percent Predicted Slow Vital Capacity
Description: Slow vital capacity measures slow and gradual expulsion of air from the lungs using a spirometer.
Time Frame: Baseline, Week 50
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of predicted volume
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 19 | 9
percentage of predicted volume | -20.9 (19.74) | -21.3 (13.90)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events, and TEAEs Leading To Study Drug Discontinuation
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or procedure, whether or not considered related to the medicinal product or procedure, which occurred during the course of the clinical study. TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 156
Population: Safety Set included all participants who received at least 1 dose of study drug grouped by treatment actually received (for reporting exposure and safety data).
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 255 | 127
Participants
  TEAEs | 204 | 108
  Treatment Emergent Serious AEs | 41 | 24
  TEAE Leading to Study Drug Discontinuation | 2 | 0

5. Secondary Outcome: Change From Baseline In Muscle Strength As Assessed By Handheld Dynamometry
Description: Handheld dynamometry (HHD) is a procedure for quantitative strength testing. Muscle strength testing was performed on prespecified muscles in the upper and lower extremities bilaterally and the force measurements were recorded. Force of measurement is reported in megascores (lower, upper, total). The total megascore is defined as the average of the non-missing ratios over baseline for all the muscles involved. The megascore at baseline is always 100. The range of a potential megascore can not be determined in advance. A megascore >100 indicates more strength compared to baseline.
Time Frame: Baseline, Week 50
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % (as the unit of megascore)
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 26 | 13
% (as the unit of megascore) | -46.5 (27.57) | -53.4 (20.28)

6. Secondary Outcome: Change From Baseline In Serum Neurofilament Light Chain
Time Frame: Baseline, Week 50
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 14 | 7
picograms/milliliter | 91.5 (40.40) | 73.1 (27.82)

7. Secondary Outcome: Change From Baseline in Serum Ravulizumab Concentration Over the Study Duration
Time Frame: Baseline, Predose at Week 50
Population: Pharmacokinetic Analysis Set (PKAS) included all participants who received at least 1 dose of the study drug and had at least 1 postdose pharmacokinetic (PK) sample. This endpoint was planned to be reported for Ravulizumab arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter
Arm/Group | Ravulizumab
Number analyzed (Participants) | 14
micrograms/milliliter | 634 (29.1)

8. Secondary Outcome: Change From Baseline in Serum Free Complement Component 5 (C5) Concentration Over the Study Duration
Time Frame: Baseline, Predose at Week 50
Population: Pharmacodynamic analysis set (PDAS) included all participants who received at least 1 dose of the study drug and had at least 1 postdose pharmacodynamics (PD) sample. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure. There were no participants with evaluable C5 data in the Placebo arm at Week 50.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 13 | 0
micrograms/milliliter | -155.2 (24.42) |

9. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADAs) to ALXN1210
Description: Blood samples were collected to evaluate antibody response through development of ADAs.
Time Frame: Week 50
Population: PDAS included all participants who received at least 1 dose of the study drug and had at least 1 postdose PD sample. Here, Number of Participants analyzed signifies those participants who were evaluable at Week 50. There were no participants with evaluable C5 data in the Placebo arm at Week 50.
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 23 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: Baseline up to Week 156
Description: Safety Set included all participants who received at least 1 dose of study drug grouped by treatment actually received (for reporting exposure and safety data). "All-Cause Mortality" reports all deaths that occurred during the study, including the deaths that led to Study Discontinuation.
Groups:
- Randomized Controlled Period: Ravulizumab: Participants received a weight-based loading dose of ravulizumab on Day 1, followed by a weight-based maintenance dose on Day 15, then q8w up to Week 42 (inclusive).
- Randomized Controlled Period: Placebo: Participants received a weight-based loading dose of placebo matched to ravulizumab on Day 1, followed by a weight-based maintenance dose on Day 15, then q8w up to Week 42 (inclusive).
- Open Label Extension Period: Ravulizumab: Participants received ravulizumab, with a blinded 900 mg dose at Week 50, followed by an open-label ravulizumab maintenance dose at Week 52, then q8w for up to 106 weeks of treatment.
- Open Label Extension Period: Placebo: Participants received ravulizumab, with a blinded loading dose at Week 50, followed by an open-label ravulizumab maintenance dose at Week 52, then q8w for up to 106 weeks of treatment.
Arm/Group | Randomized Controlled Period: Ravulizumab | Randomized Controlled Period: Placebo | Open Label Extension Period: Ravulizumab | Open Label Extension Period: Placebo
All-Cause Mortality (participants affected / at risk) | 15/255 | 6/127 | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 41/255 | 24/127 | 2/14 | 0/5
Other Adverse Events (participants affected / at risk) | 196/255 | 106/127 | 3/14 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Controlled Period: Ravulizumab (N=255) | Randomized Controlled Period: Placebo (N=127) | Open Label Extension Period: Ravulizumab (N=14) | Open Label Extension Period: Placebo (N=5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Assisted suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeding tube user (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Controlled Period: Ravulizumab (N=255) | Randomized Controlled Period: Placebo (N=127) | Open Label Extension Period: Ravulizumab (N=14) | Open Label Extension Period: Placebo (N=5)
Fall (Injury, poisoning and procedural complications) | 54 (81) | 36 (65) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 11 (13) | 8 (13) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 26 (29) | 5 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (28) | 10 (10) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 9 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 42 (62) | 22 (29) | 1 (1) | 0 (0)
Fatigue (General disorders) | 22 (40) | 11 (11) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 21 (31) | 5 (7) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (23) | 4 (5) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (12) | 11 (12) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 13 (14) | 8 (8) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The IDMC recommended the study be discontinued due to lack of efficacy with ravulizumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT04248465/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT04248465/SAP_001.pdf